CLINICAL TRIAL: NCT05304572
Title: Interobserver Agreement of Determination of Hepatocellular Carcinoma Feeding Vessels : Multi-Detector CT Angiography With 3D Reconstruction Versus Digital Subtraction Angiography
Brief Title: Multi-Detector CT Angiography With 3D Reconstruction Versus Digital Subtraction Angiography
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy Mohammed Ahmed, lecturer of interventional and diagnostic radiology, Assiut University
Other Study IDs: MDCT angiography HCC
Record Dates: First submitted 2022-02-04; First posted 2022-03-31 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Three-Dimensional CT Angiography; HCC; TACE; DSA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multi-Detector CT angiography — Multiphasic CT within 4 weeks interval prior to TACE will be done including non-enhanced, arterial, portal and venous phases using IV bolus injection of a 75-100-mLiodinated contrast material iopamidol at a rate of 3.0 mL/s. The images of arterial phase will be transferred to workstation to produce 3D angiographic reconstruction images .
Procedure: Trans-arterial chemoembolization and DSA — Percutaneous arterial access is achieved through the common femoral artery (19 G needle) under local anesthesia with placement of a 5-Fr sheath. A 5-Fr Cobra (C2) or sidewinder (SIM1) catheter was used for catheterizing the coeliac trunk and SMA. Then celiac and superior mesenteric angiography was done by injecting 24 mL of iopamidol using forced manual injection method or using a pump at a rate of 6 mL/s according to the operator preferences.Then a microcatheter was used for selective and super-selective access of the hepatic arteries. The micro-catheter was placed in the feeding artery as close as possible to the tumor.The chemotherapeutic drugs (Doxorubicin 50 mg) solved within 5 ml of iodinated non-ionic contrast media and then mixed with 10 ml of iodized oil (lipiodol) will be delivered through the feeding hepatic artery and then embolized using Poly-vinyl Alcohol (PVA) particles.

SUMMARY:
This study aims to investigate the feasibility and accuracy of Multi-Detector CT angiography acquired before Trans-arterial Chemo-embolization (TACE) in detecting Hepato-cellular carcinoma feeding vessels compared to DSA angiography acquired during TACE.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) represents the sixth most common cancer worldwide. Trans-arterial chemoembolization (TACE) is a palliative treatment for patients with HCC who are not candidates for transplantation, surgical resection, or loco-regional ablation. This minimally invasive procedure allows delivery of a high concentration of particles and/or chemotherapeutic agents into the liver, causing ischemic cell death and permitting local delivery of high concentrations of chemotherapeutic drug. Selective administration of chemo-embolic material to the tumor is desired, where possible, to increase the effectiveness of treatment to the tumor and minimize injury to surrounding liver tissue.

Tumor detection and assessment of the tumor-feeding vessel(s) are important for an effective treatment, while limiting non-target embolization. Usually, selection of the tumor-feeding vessels during TACE has been guided by 2D digital subtraction angiography (DSA). However; this method has a disadvantage of occasional misinterpretation of tumor-feeding vessels due to superimposition of vessels. To prevent such misinterpretation, multiple selective injections and oblique projections are performed during TACE with consequent increase in procedure time, volume of injected contrast material, and radiation doses.

A relatively new approach using three-dimensional (3D) cone-beam CT angiography during TACE is reported to be extremely helpful, especially in cases of complex hepatic arterial anatomy. However, the time required for processing and evaluating this 3D angiography images may discourage its routine use by intervention radiologists because it requires either a sterile remote control for in-room review or the operator exit from the angiographic room to access a workstation. A new automatic specifically designed softwares has been developed for detection of feeding vessels after Cone beam CT, but these softwares are not widely available.

Multiphasic contrast enhanced CT is one of the recommended imaging tools for diagnosis of HCC and is routinely done before TACE. There are few reports on the application of Multi-Detector CT angiography for detection of HCC feeding vessels before TACE.

This study aims to investigate the feasibility and accuracy of Multi-Detector CT angiography for assessment of tumor-feeding vessel in patients planned for TACE compared to DSA angiography acquired during TACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC not suitable for resection, liver transplantation, or percutaneous ablation.
* CHILD class A/B cirrhosis.
* patent main portal vein.
* less than 50% involvement of the liver by the tumor.
* no vascular invasion or extrahepatic spread of the HCC.
* normal renal functions.
* bilirubin level < 2 mg/dl .

Exclusion Criteria:

* Pre-TACE Multi-Detector CT raw DICOM images could not be obtained for 3D processing
* patients with only available Pre-TACE MRI images
* Failed TACE due to technical factors
* Non-selective TACE technique

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 70 consecuetive patients referred for TACE after evaluation by the multidisciplinary team at our hospital according to Barcelona clinic liver cancer (BCLC) classification and recommended treatment options.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
feeding vessels detectability | Baseline
  The observers will evaluate DSA images of the celiac, superior mesenteric artery (SMA), common hepatic artery (CHA), right or left hepatic arteries obtained during TACE and record possible feeding arteries. Observers will be blind to additional angio-grams obtained during TACE i.e selective DSA images of the segmental arteries and feeding arteries. observers will then evaluate the CT 3D images and record possible feeding arteries. The ''ground truth'' (GT) will be the gold standard tool and is obtained after completing the above mentioned analyses by allowing the observers to evaluate by consensus pre-embolization CT 2D and 3D images, all acquired DSA images during TACE , and post-lipiodol injection CT images if available. GT was used to define true-positive, false-positive, false-negative and true negative feeding vessels.

SECONDARY OUTCOMES:
inter-observer agreement | Baseline
  Interobserver variability was assessed using kappa statistics. Interobserver agreement was defined as excellent, fair to good, and poor by kappa values of >0.75, 0.40-0.75, and <0.40, respectively. for each technique.

CONTACTS AND LOCATIONS:
Overall Officials: Ramy M Ahmed, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut Universtiy Hospital; Alrajhy Liver institute, Asyut, Egypt

REFERENCES:
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Brown DB, Geschwind JF, Soulen MC, Millward SF, Sacks D. Society of Interventional Radiology position statement on chemoembolization of hepatic malignancies. J Vasc Interv Radiol. 2009 Jul;20(7 Suppl):S317-23. doi: 10.1016/j.jvir.2009.04.015. No abstract available. PMID 19560017
- [Background] Marelli L, Stigliano R, Triantos C, Senzolo M, Cholongitas E, Davies N, Tibballs J, Meyer T, Patch DW, Burroughs AK. Transarterial therapy for hepatocellular carcinoma: which technique is more effective? A systematic review of cohort and randomized studies. Cardiovasc Intervent Radiol. 2007 Jan-Feb;30(1):6-25. doi: 10.1007/s00270-006-0062-3. PMID 17103105
- [Background] Liapi E, Hong K, Georgiades CS, Geschwind JF. Three-dimensional rotational angiography: introduction of an adjunctive tool for successful transarterial chemoembolization. J Vasc Interv Radiol. 2005 Sep;16(9):1241-5. doi: 10.1097/01.RVI.0000174283.03032.8E. PMID 16151066
- [Background] Kakeda S, Korogi Y, Ohnari N, Moriya J, Oda N, Nishino K, Miyamoto W. Usefulness of cone-beam volume CT with flat panel detectors in conjunction with catheter angiography for transcatheter arterial embolization. J Vasc Interv Radiol. 2007 Dec;18(12):1508-16. doi: 10.1016/j.jvir.2007.08.003. PMID 18057285
- [Background] Miyayama S, Yamashiro M, Okuda M, Yoshie Y, Sugimori N, Igarashi S, Nakashima Y, Matsui O. Usefulness of cone-beam computed tomography during ultraselective transcatheter arterial chemoembolization for small hepatocellular carcinomas that cannot be demonstrated on angiography. Cardiovasc Intervent Radiol. 2009 Mar;32(2):255-64. doi: 10.1007/s00270-008-9468-4. Epub 2008 Dec 9. PMID 19067043
- [Background] Chiaradia M, Izamis ML, Radaelli A, Prevoo W, Maleux G, Schlachter T, Mayer J, Luciani A, Kobeiter H, Tacher V. Sensitivity and Reproducibility of Automated Feeding Artery Detection Software during Transarterial Chemoembolization of Hepatocellular Carcinoma. J Vasc Interv Radiol. 2018 Mar;29(3):425-431. doi: 10.1016/j.jvir.2017.10.025. Epub 2018 Feb 3. PMID 29402612
- [Background] Deschamps F, Solomon SB, Thornton RH, Rao P, Hakime A, Kuoch V, de Baere T. Computed analysis of three-dimensional cone-beam computed tomography angiography for determination of tumor-feeding vessels during chemoembolization of liver tumor: a pilot study. Cardiovasc Intervent Radiol. 2010 Dec;33(6):1235-42. doi: 10.1007/s00270-010-9846-6. PMID 20390271
- [Background] Bruix J, Sherman M, Llovet JM, Beaugrand M, Lencioni R, Burroughs AK, Christensen E, Pagliaro L, Colombo M, Rodes J; EASL Panel of Experts on HCC. Clinical management of hepatocellular carcinoma. Conclusions of the Barcelona-2000 EASL conference. European Association for the Study of the Liver. J Hepatol. 2001 Sep;35(3):421-30. doi: 10.1016/s0168-8278(01)00130-1. No abstract available. PMID 11592607
- [Background] Huang JH, Fan WJ, Li CJ, Gu YK, Zhang L, Gao F, Lu LW, Li WQ. Application of multislice spiral CT angiography on transcatheter arterial chemoembolization for hepatocellular carcinoma. Ai Zheng. 2009 Feb;28(2):159-63. Epub 2009 Feb 15. PMID 19550129
- [Background] Kim I, Kim DJ, Kim KA, Yoon SW, Lee JT. Feasibility of MDCT angiography for determination of tumor-feeding vessels in chemoembolization of hepatocellular carcinoma. J Comput Assist Tomogr. 2014 Sep-Oct;38(5):742-6. doi: 10.1097/RCT.0000000000000103. PMID 24834885
- [Derived] Ahmed RM, Ali WA, AbdelHakam AM, Ahmed SH. Detection of hepatocellular carcinoma feeding vessels: MDCT angiography with 3D reconstruction versus digital subtraction angiography. BMC Med Imaging. 2024 Sep 18;24(1):250. doi: 10.1186/s12880-024-01408-z. PMID 39294600